CLINICAL TRIAL: NCT05703425
Title: The Effect of Sulfasalazine on CRH Levels in Pregnant Women With a History of Pre-Term Birth: A Randomized Controlled Trial
Brief Title: The Effect of Sulfasalazine on CRH Levels in Pregnant Women
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Emily B. Rosenfeld, DO, RBHS Instructor, Divisions of Maternal-Fetal Medicine, and Epidemiology and Biostatistics, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro2021001951
Record Dates: First submitted 2023-01-17; First posted 2023-01-30 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Preterm Birth
Keywords: preterm birth; sulfasalazine; corticotropin releasing hormone; randomized controlled trial
MeSH Terms: conditions — Premature Birth | interventions — Sulfasalazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sulfasalazine (Experimental): Pregnant persons will receive sulfasalazine daily with 500 mg/daily and increasing by 500 mg/day every week until they reach a therapeutic dose of 1,000 mg twice daily. Drug will be started at 24 weeks estimated gestational age and ended at 36 weeks or earlier if preterm birth occurs.
  Interventions: Drug: Sulfasalazine
- Standard Care (No Intervention): Pregnant persons will receive standard care in pregnancy.

INTERVENTIONS:
Drug: Sulfasalazine — Sulfasalazine will be administered between 24 and 36 weeks of pregnancy
  Arms: Sulfasalazine

SUMMARY:
The goal of this randomized clinical trial is to assess sulfasalazine as a potential treatment to prevent recurrent preterm birth. The main questions it aims to answer are:

* Does sulfasalazine down regulate corticotropin releasing hormone (CRH) levels in pregnant persons with a prior history of preterm birth?
* Does sulfasalazine reduce the incidence of recurrent preterm birth in pregnant persons given drug vs. controls?

Consenting participants will be randomized to receive sulfasalazine or to a control group and will undergo serial blood draws to assess plasma CRH levels.

DETAILED DESCRIPTION:
This is a study to assess the potential for sulfasalazine to prevent recurrent preterm birth. The investigators' main objective is to assess the effects of sulfasalazine on the maternal serum biomarker CRH, which is associated with preterm birth.

The will be a pilot randomized controlled trial of pregnant multiparous patients who have had a prior preterm delivery. Pregnant women with a prior preterm birth are at high risk (about 20-30%) of having a recurrent preterm birth. The goal of the study will be to evaluate the effect of sulfasalazine on the maternal serum biomarker CRH at 28, 32, and 36 weeks gestation after randomization of patients to the study drug.

Secondary objectives include evaluating the effect of sulfasalazine on the outcome of delivery less than 37 weeks gestation in this group of high risk pregnant women. Additional composite neonatal outcomes will be assessed.

The proposed study has the potential to identify a novel, low-cost, orally available treatment for preterm delivery based on in vitro evidence and epidemiologic studies suggesting that sulfasalazine may be an effective intervention to prevent preterm birth. If the hypothesis put forth by the investigators is confirmed, sulfasalazine would be an attractive therapeutic intervention that could be implemented for the prevention of preterm birth in both developed and developing nations.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years of age
* Singleton pregnancy
* Participants with a history of prior preterm birth in a previous pregnancy
* Participants must be between 12 and 22 weeks gestation.
* Participants must have their pregnancy dates confirmed by ultrasound.

Exclusion Criteria:

* Participants < 18 years old
* Participants with a cervical length < 25 mm
* Participants with a multiple gestation
* Cerclage
* Progesterone administration
* Unwilling or unable to swallow the study agent capsule or consume an inert ingredient in the study agent capsule
* Acute liver disease or known liver abnormalities
* Other significant chronic medical or psychiatric illness that, in the investigator's opinion, would prevent participation in the study
* Known hypersensitivity to sulfasalazine
* Known glucose-6-phosphate dehydrogenase (G6PD) deficiency
* History of severe asthma
* Digoxin use
* Porphyria
* Intestinal obstruction
* Urinary tract obstruction
* Hepatic dysfunction
* Renal dysfunction
* Blood dyscrasia such as agranulocytosis, aplastic anemia.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Serum CRH levels | between 28 and 36 weeks of pregnancy
  CRH will be assessed at 28, 32, and 36 weeks gestation

SECONDARY OUTCOMES:
Spontaneous preterm birth < 37 weeks gestation | up to 37 weeks of pregnancy
  Preterm births prior to 37 weeks secondary to preterm labor (PTL) or premature Preterm births secondary to preterm labor or preterm rupture of the membranes (PPROM)
Spontaneous preterm birth < 34 weeks gestation | up to 34 weeks of pregnancy
  Preterm births prior to 34 weeks secondary to PTL or PPROM
Medically indicated preterm birth < 37 weeks gestation | up to 37 weeks of pregnancy
  Preterm births due to maternal or fetal disease not related to PTL or PPROM
Digital cervical exam at 36 weeks gestational age | between 35 weeks and 36 weeks 6 days of pregnancy
  Digital cervical exam at 36 weeks gestational age
Composite neonatal morbidity | From birth of the neonate until 28 days of life
  Composite outcome including but not limited to Apgar neonatal death, respiratory distress, necrotizing enterocolitis, and bronchopulmonary dysplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Rosenfeld, DO, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be provided to those inquire to the corresponding author of the manuscript if published. If no manuscript is published, inquiries can be directed to the principal investigator of the study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available on publication and remain available for two years.
Access Criteria: The principal investigator will individually assess all requests for data.

REFERENCES:
- [Background] McLean M, Bisits A, Davies J, Woods R, Lowry P, Smith R. A placental clock controlling the length of human pregnancy. Nat Med. 1995 May;1(5):460-3. doi: 10.1038/nm0595-460. PMID 7585095
- [Background] Wang B, Parobchak N, Rosen T. RelB/NF-kappaB2 regulates corticotropin-releasing hormone in the human placenta. Mol Endocrinol. 2012 Aug;26(8):1356-69. doi: 10.1210/me.2012-1035. Epub 2012 Jun 25. PMID 22734038
- [Background] Wang B, Parobchak N, Martin A, Rosen M, Yu LJ, Nguyen M, Gololobova K, Rosen T. Screening a small molecule library to identify inhibitors of NF-kappaB inducing kinase and pro-labor genes in human placenta. Sci Rep. 2018 Jan 26;8(1):1657. doi: 10.1038/s41598-018-20147-0. PMID 29374256
- [Background] Norgard B, Fonager K, Pedersen L, Jacobsen BA, Sorensen HT. Birth outcome in women exposed to 5-aminosalicylic acid during pregnancy: a Danish cohort study. Gut. 2003 Feb;52(2):243-7. doi: 10.1136/gut.52.2.243. PMID 12524407
- [Background] Mogadam M, Dobbins WO 3rd, Korelitz BI, Ahmed SW. Pregnancy in inflammatory bowel disease: effect of sulfasalazine and corticosteroids on fetal outcome. Gastroenterology. 1981 Jan;80(1):72-6. PMID 6108894
- [Background] Hensleigh PA, Kauffman RE. Maternal absorption and placental transfer of sulfasalazine. Am J Obstet Gynecol. 1977 Feb 15;127(4):443-4. doi: 10.1016/0002-9378(77)90510-5. No abstract available. PMID 13655